CLINICAL TRIAL: NCT07043959
Title: Comparative Effects of Isometrics Versus Range of Motion Exercises on Pain, Mobility and Functional Independence in Post-Mastectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Dr Izza Ayub; PT, Principal Investigator, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/PB/40/1033/40
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: Post Mastectomy; Postmastectomy Pain
Keywords: Isometric Exercises; Range of Motion Exercises; Pain; Mobility; Functional Independence; Post-mastectomy
MeSH Terms: conditions — Pain | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometrics Exercise Group A (Experimental): Group A received a hot pack for 10-15 minutes and performed deep breathing exercises for 3-4 repetitions. Patients were instructed in diaphragmatic breathing, where they inhaled deeply, held their breath for 2-3 seconds, and then exhaled. Following this, isometric exercises were performed, consisting of 2 sets of each exercise with 5-7 repetitions per set, done three times per week for a total duration of 8 weeks.
  Interventions: Procedure: Isometrics Exercise
- Range of Motion Exerccise Group B (Active Comparator): Group B received a hot pack for 10-15 minutes and performed deep breathing exercises for 3-4 repetitions. Patients were guided in diaphragmatic breathing, where they inhaled deeply, held their breath for 2-3 seconds, and then exhaled. Afterward, they performed Range of Motion (ROM) exercises, consisting of 2 sets of each exercise with 5-7 repetitions per set, conducted three times per week over a period of 8 weeks.
  Interventions: Procedure: Range of Motion Exercises

INTERVENTIONS:
Procedure: Isometrics Exercise — Shoulder Squeeze:
  The therapist instructed the patient to lift their arms to shoulder height while keeping the elbows bent, then move the arms backward until the shoulder blades come together.
  Arm Lift to Front and Side:
  The therapist instructed the patient to raise their arm forward and upward while applying gentle resistance for 2-3 seconds to facilitate front arm elevation. Then, the patient was guided to lift the arm sideways, with slight resistance applied for 2-3 seconds to assist in side-arm elevation.
  Arms: Isometrics Exercise Group A
Procedure: Range of Motion Exercises — Wall Climb for Flexion: The therapist instructed the patient to move their fingers upward along the wall until they reach their limit, then repeat the movement.
  Arm across Chest for Adduction and Internal Rotation: The therapist instructed the patient to move the affected arm toward the unaffected arm and shoulder.
  Wand Exercise for Flexion and Abduction: The patient was instructed to hold a wand with both hands and move it forward and sideways toward the affected side
  Arms: Range of Motion Exerccise Group B

SUMMARY:
The aim of study was to investigate the comparative effectiveness of Isometrics versus Range of Motion (ROM) Exercises on Pain, Mobility and Functional Independence post-mastectomy. A randomized clinical trial was conducted, in which 30 participants were randomly assigned to 2 parallel groups. One group received Isometric Exercises, while the other received Range of Motion Exercises. Outcome measures included pain, range of motion and functional independence. Treatments were administered 3 times per week with 2 sets of each exercise with 5-7 repetitions per day for a duration of eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 45 and 65
* Underwent a one-sided mastectomy
* No history of shoulder injuries
* Able to understand instructions and provide informed consent

Exclusion Criteria:

* Experiencing severe pain
* Diagnosed with advanced lymph edema
* Physically unable to engage in exercises
* Medically unstable

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 30 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain | Eight Weeks
  Numeric Pain Rating Scale (NPRS) with decreasing values indicates improved patient condition and reduced pain intensity.
Shoulder ROM | Eight Weeks
  Goniometer with increasing ROM indicates improved patient condition and joint movements.

SECONDARY OUTCOMES:
Shoulder Functional Independence | Eight Weeks
  Upper Extremity Functional Scale determines the level of function of participant where higher score indicates improved upper extremity function and reduced functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Izza Ayub; PT, Principal Investigator — Department of Rehabilitaion Sciences, The University of Faisalabad
Locations (1):
- The University of Faisalabad, Faisalābad, Pakistan